CLINICAL TRIAL: NCT04805424
Title: Different Techniques for Abdominoplasty After Massive Weight Loss: Safety and Outcomes
Brief Title: Techniques for Abdominoplasty After Massive Weight Loss
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Karolinska University Hospital unable to support the clinical trial as anticipated.
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Ebba Lindqvist, Principal Investigator, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-06151
Record Dates: First submitted 2021-03-10; First posted 2021-03-18 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Skin; Excess
Keywords: Randomized controlled trial; Abdominoplasty; Massive weight loss; Plastic surgery; Liposuction
MeSH Terms: interventions — Abdominoplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominoplasty (Active Comparator): Standard abdominoplasty
  Interventions: Procedure: Abdominoplasty
- Lipo-abdominoplasty (Experimental): Abdominoplasty plus liposuction
  Interventions: Procedure: Lipo-abdominoplasty

INTERVENTIONS:
Procedure: Lipo-abdominoplasty — Abdominoplasty plus liposuction
  Arms: Lipo-abdominoplasty
Procedure: Abdominoplasty — Abdominoplasty
  Arms: Abdominoplasty

SUMMARY:
Excess skin on the abdomen is a common problem for many individuals after massive weight loss. The surgical procedure of abdominoplasty is intended to remove excess skin and improve the shape of the torso in abdomen, in order to address issues such as skin fold eczema, difficulties finding clothing, and psychosocial issues.

The investigators will conduct a randomized, controlled trial where individuals with excess skin on the abdomen will be randomized to either standard abdominoplasty or abdominoplasty in combination with liposuction. The investigators will examine the rate of complications, and the functional and aesthetical outcomes of the two methods.

ELIGIBILITY:
This study is open only to individuals who are residents in Sweden and qualify for government-funded, inpatient, non-emergency health care within the Stockholm Region.

Inclusion Criteria:

* BMI < 30
* Stable BMI for >= 6 months
* >= 24 months since bariatric surgery, if applicable
* Skin fold of >= 5 cm
* Functional and/or psychosocial issues due to abdominal skin excess

Exclusion Criteria:

* Smoking
* Ongoing infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of and type of complications within 30 days | 30 days
  Number of and type of complications occurring within 30 days of surgery

SECONDARY OUTCOMES:
Average need for analgesia in morphine equivalents | Post-operative day 1
  Average need for analgesia in morphine equivalents during post-operative day 1
Average score on BodyQ score | At baseline, at 3 months post-operatively, at 12 months post-operatively
  Average score on BodyQ score including subscales. BodyQ is developed and owned by Memorial Sloan Kettering Cancer Center. The BODY-Q is composed of 27 independently functioning scales that measure 3 overarching constructs Appearance, Quality of Life and Experience of Care. Scales are translated to a 0-100 score where a lower score means worse outcome.
Average score on aesthetic result | At 12 months post-operatively
  Average score on aesthetic result on a 1-10 scale where a lower score means worse outcome.
Average days until discharge | Days
  Average days until discharge post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Ebba Lindqvist, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Reconstructive Plastic Surgery, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No